CLINICAL TRIAL: NCT00539604
Title: Phase IV Multicenter, Intra-Individually Controlled, Comparison Study to Evaluate the Negative Predictive Value of 16-64 Slice MDCT Imaging in Patients Scheduled for Coronary Angiography
Brief Title: Non Invasive Multicenter Italian Study for Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Società Italiana di Radiologia Medica (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMIS-CAD
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2006-11

CONDITIONS: Coronary Heart Disease
Keywords: Comparison study between MDCT and coronary angiography
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Procedure: MDCT and Coronary Angiography

SUMMARY:
To determine if 16-64 slice multidetector CT (MDCT) can replace the invasive procedure in patients scheduled for coronary angiography in order to exclude the presence of CAD

DETAILED DESCRIPTION:
Because coronary artery disease (CAD) is the most frequent cause of death in industrialized nations and its onset is currently unpredictable, there is a need for new methods of screening apparently healthy individuals to identify those at increased risk.

Several imaging techniques are in use to visualize coronary arteries. These include both invasive procedure as x-ray coronary angiography and those non invasive like computed tomography (CT) and magnetic resonance imaging (MRI). Among these imaging modalities, selective cardiac catheterization and x-ray angiography is the current gold standard for visualization of coronaries and detection of their stenoses, providing for optimal spatial resolution, a general "road map" of the coronary tree for interventions. The replacement of even a fraction of these procedures with non-invasive modalities would constitute an important advance in the care of patients with suspected coronary artery disease Preliminary results reported in literature addressing the study of coronary arteries by multidetector-CT (MDCT) appear to be interesting. Several studies have been performed firstly using Electron beam CT (EBCT).EBCT provides high temporal resolution and enables quantitative assessment of the coronary artery calcium, but because of limited spatial resolution as a result of limited z axis resolution, it does not permit direct visualisation in multi-reformation of the whole coronary artery system.

With the introduction of 4-row MDCT there have now been several studies aimed to compare the MDCT with a standard invasive angiography. Data published for over 200 subjects from 4 studies demonstrated that patient compliance at breath-hold, heart rate and rhythm are crucial limitation to this procedure. In the Nieman and Achembach papers not all the coronary segments were assessable because of the limited temporal resolution of 4-slice MDCT. With this machine it is mandatory to select patients carefully, considering only those with baseline hearth rate < 65 bpm (also obtained by pre-treatment with β-blockers in order to slow hearth rate).

ELIGIBILITY:
Inclusion Criteria:

1. Patients (men or women of any ethnic group) scheduled for a coronary angiography evaluation for a diagnostic work up.
2. Patients will be expected to undergo coronary angiography within 2 weeks after the MDCT study procedure. The coronary angiography must meet the minimum standard laid down in the protocol (see section 8.3.3).
3. Patients must have HDL and total cholesterol performed within the last year.
4. Patients must be willing and able to continue study participation following the reference test to ensure completion of all procedures and observations required by the study.
5. Fully informed and signed consent must be obtained from each patient.

   -

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patients who have received any investigational drug within the 30 days prior to entering this study.
3. Pregnant or lactating women.
4. Patients who have any contraindication to MDCT examination with iodinate contrast media.
5. Patients with heart rate >70 bpm despite of β-blocker treatment (see section 8.2.4.1).
6. Patients with no sinus rhythm.
7. Patients with NYHA III or IV class.
8. Patients who have previously undergone CABG or stenting.
9. Patients with a creatinine value > 2 mg/dl.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2004-07; Study Completion 2006-06

PRIMARY OUTCOMES:
to determine if 16-64 slice multidetector CT (MDCT) can replace the invasive procedure in patients scheduled for coronary angiography in order to exclude the presence of CAD

SECONDARY OUTCOMES:
the efficacy in terms of performance of the MDCT in each single coronary segment and
the safety in terms of AE related to both procedures

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Del Maschio, Med. Doctor, Principal Investigator; Lorenzo Bonomo, Med. Doctor, Principal Investigator
Locations (20):
- Italy (20):
  - Policlinico di Bari Istituto di Radiologia, Bari, Ba
  - Policlinico S. Orsola Malpighi Istituto di Radiologia III, Bologna, Bo
  - Azienda Istituti Ospitalieri U.O. Radiologia, Cremona, CR
  - Istituti clinici Humanitas, Rozzano, Milano
  - Ospedale San Raffaele Istituto di Radiologia, Milan, MI
  - Centro Cardiologico Monzino Servizio di Radiologia, Milan, MI
  - Policlinico di Modena Istituto di Radiologia, Modena, Mo
  - Ospedale G. Pasquinucci Unità Operativa di Radiologia, Massa, Ms
  - Policlinico P. Giaccone Dip. Scienze Radiologiche, Palermo, Pa
  - A.O. Riuniti Unità Operativa di Radiologia, Reggio Calabria, R.C.
  - Policlinico Le Scotte DAI dell' Immagine, Siena, SI
  - A.O. S. Maria Dipartimento di Diagnostica per Immagini, Terni, TN
  - Ospedale S. Chiara Dipartimento di Radiologia, Trento, TN
  - Ospedale Molinette Istituto di Radiologia, Torino, To
  - Ospedale S. Maria di Ca' Foncello U.C. Radiologia, Treviso, TV
  - A.O.R.N. Cardarelli Radiologia Generale I Sez., Napoli
  - Policlinico Tor Vergata Istituto di Radiologia, Roma
  - Policlinico Umberto I Radiologia D.E.A., Roma
  - Policlinico Umberto I Università degli Studi "La Sapienza" Dip. Scienze Radiologiche, Roma
  - Policlinico Gemelli Istituto di Radiologia, Roma